CLINICAL TRIAL: NCT02246335
Title: Hemiarthroplasty Compared to Total Hip Arthroplasty for Displaced Femoral Neck Fractures in the Elderly-elderly. A Randomized Controlled Trial.
Brief Title: Hemiarthroplasty Compared to Total Hip Arthroplasty for Displaced Femoral Neck Fractures in the Elderly-elderly
Acronym: HOPE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Danderyd Hospital (Other)
Responsible Party: Principal Investigator, Olof Skoldenberg, Medical Doctor, Ph D, Danderyd Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HOPE
Record Dates: First submitted 2014-09-18; First posted 2014-09-22 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Femoral Neck Fractures
MeSH Terms: conditions — Femoral Neck Fractures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (Active Comparator): Hemiarthroplasty
  Interventions: Device: Cemented hemiarthroplasty
- Treatment group (Active Comparator): Total hip arthroplasty
  Interventions: Device: Cemented total hip arthroplasty

INTERVENTIONS:
Device: Cemented total hip arthroplasty
  Arms: Treatment group
Device: Cemented hemiarthroplasty
  Arms: Control group

SUMMARY:
Total Hip Arthroplasty is equal to or better than Hemiarthroplasty in the treatment of displaced femoral neck fractures in the elderly-elderly

DETAILED DESCRIPTION:
Total Hip Arthroplasty is equal to or better alternative to Hemiarthroplasty in the treatment of displaced femoral neck fractures in the elderly-elderly (patients 80 years and over).

ELIGIBILITY:
Inclusion Criteria:

* Acute displaced femoral neck fracture of hip (Garden classification 3-4)
* Independent walker with or without walking aides
* Patient willing to participate in the study and give written consent.

Exclusion Criteria:

* Fracture older than 36 hours before admission
* Osteoarthritis in the fractured hip
* Rheumatoid arthritis in the fractured hip
* Pathological fractures
* Contraindication for hip arthroplasty surgery
* Not suitable for inclusion for other reasons e.g. substance abuse

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-10; Primary Completion 2016-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Harris hip score | 2 years
  The hip specific outcome score Harris hip score at 2 years will be the main outcome variable

SECONDARY OUTCOMES:
EQ-5D | 2 years
  Health-related quality of life at 2 years
EQ-5D | 4 years
  Health-related quality of life at 4 years
EQ-5D | 6 years
  Health-related quality of life at 6 years
EQ-5D | 10 years
  Health-related quality of life at 10 years
Adverse events | 2 years
  All hip related adverse events at 2 years
Adverse events | 4 years
  All hip related adverse events at 4 years
Adverse events | 6 years
  All hip related adverse events at 6 years
Adverse events | 10 years
  All hip related adverse events at 10 years
Harris hip score | 4 years
  Harris hip score at 4 years
Harris hip score | 6 years
  Harris hip score at 6 years
Harris hip score | 10 years
  Harris hip score at 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- Orthopaedic department, Danderyd Hospital, Stockholm, Stockholm County, Sweden

REFERENCES:
- [Derived] Skoldenberg O, Chammout G, Mukka S, Muren O, Nasell H, Hedbeck CJ, Salemyr M. HOPE-trial: hemiarthroplasty compared to total hip arthroplasty for displaced femoral neck fractures in the elderly-elderly, a randomized controlled trial. BMC Musculoskelet Disord. 2015 Oct 19;16:307. doi: 10.1186/s12891-015-0763-3. PMID 26480938